CLINICAL TRIAL: NCT06046586
Title: Randomized Factorial Trial of Internet-Delivered Psychological Treatment for Cancer Survivors With Clinically Significant Psychiatric Symptoms
Brief Title: Internet-Delivered Psychological Treatment for Cancer Survivors
Acronym: IN-FACT-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erland Axelsson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04056-01 #2
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cancer Survivors; Anxiety; Depression
Keywords: psycho-oncology; randomized factorial trial; Internet-delivered cognitive behavior therapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Internet-delivered psychological treatment, arm #1 (Experimental): Support and information + Behavioral activation
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation
- Internet-delivered psychological treatment, arm #2 (Experimental): Support and information + Systematic exposure with mindfulness training
  Interventions: Behavioral: Support and information; Behavioral: Systematic exposure with mindfulness training
- Internet-delivered psychological treatment, arm #3 (Experimental): Support and information + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #4 (Experimental): Support and information + Behavioral activation + Systematic exposure with mindfulness training
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Systematic exposure with mindfulness training
- Internet-delivered psychological treatment, arm #5 (Experimental): Support and information + Behavioral activation + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #6 (Experimental): Support and information + Systematic exposure with mindfulness training + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Systematic exposure with mindfulness training; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #7 (Experimental): Support and information + Behavioral activation + Systematic exposure with mindfulness training + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Systematic exposure with mindfulness training; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #8 (Experimental): Support and information
  Interventions: Behavioral: Support and information

INTERVENTIONS:
Behavioral: Support and information — Emotional and technical support. Information about the long-term effects of cancer.
Behavioral: Behavioral activation — Behavioral activation with existential themes and emphasis on values and relationships.
  Arms: Internet-delivered psychological treatment, arm #1; Internet-delivered psychological treatment, arm #4; Internet-delivered psychological treatment, arm #5; Internet-delivered psychological treatment, arm #7
Behavioral: Systematic exposure with mindfulness training — Systematic exposure with mindfulness training with a focus on anxiety about health and/or death, body image, and cancer-related trauma.
  Arms: Internet-delivered psychological treatment, arm #2; Internet-delivered psychological treatment, arm #4; Internet-delivered psychological treatment, arm #6; Internet-delivered psychological treatment, arm #7
Behavioral: Promotion of health behaviors — An overview of self-management techniques in terms of physical exercise, dietary advice, and strategies for improved sleep.
  Arms: Internet-delivered psychological treatment, arm #3; Internet-delivered psychological treatment, arm #5; Internet-delivered psychological treatment, arm #6; Internet-delivered psychological treatment, arm #7

SUMMARY:
Negative psychological effects of cancer are common, but cancer survivors are rarely offered structured psychological treatment. Internet-delivered treatments have shown some promise, but specific treatment components have not been empirically evaluated which means that it is not clear which therapies that should be prioritized. In this randomized factorial trial at Karolinska Institutet, Stockholm, Sweden, 400 cancer survivors with psychiatric symptoms are enrolled in variations on a 10-week therapist-guided online psychological treatment intended to address the negative psychological long-term effects of cancer. The aim is to determine the contribution of treatment components to the overall effect.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor at least 0.5 years after main therapy
* Clinically significant anxiety or depression (Patient Health Questionnaire 9 [PHQ-9]≥10, or Generalized Anxiety Disorder 7 [GAD-7]≥8, or 9-item Fear of Cancer Recurrence Inventory [FCRI-9]≥16)
* At least 18 years old
* Resident of Region Stockholms, Västra Götalandsregionen, or Region Skåne, Sweden (listed and de facto)
* Sufficient technical knowledge and knowledge of the Swedish language to take part in a text-based online treatment
* Continuous access to an electronic device that can be used to access the study web platform

Exclusion Criteria:

* Recurrent thoughts of suicide, as based on clinical judgement aided by the structured interview and the self-report version of the Montgomery-Åsberg Depression Rating Scale (MADRS-S) item 9
* Severe medical condition (e.g., very poor prognosis, stage IV cancer), severe psychiatric disorder (e.g., psychotic disorder, bipolar disorder, or severely debilitating substance use disorder, severe depression), or medical treatment (e.g., chemotherapy, immunotherapy, radiotherapy) that makes the treatment unfeasible
* Other ongoing psychological treatment
* Continuous psychotropic medication not stable for the past 4 weeks, or not expected to remain stable during the treatment period
* Planned absence for more than one week of the intended treatment period
* No complete the pre-treatment assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
General anxiety | Pre-treatment (within 2 weeks before treatment), via weekly assessments, to post-treatment (after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  General Anxiety Disorder 7 (GAD-7, theoretical range: 0-21, where a higher score indicates more general anxiety). The phrasing is revised to concern the past week. The conventional version is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Depressive symptoms | Pre-treatment (within 2 weeks before treatment), via weekly assessments, to post-treatment (after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  Patient Health Questionnaire 9 (PHQ-9, theoretical range: 0-27, where a higher score indicates more symptoms of depression). The phrasing is revised to concern the past week. The conventional version is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Fear of cancer recurrence | Pre-treatment (within 2 weeks before treatment), via weekly assessments, to post-treatment (after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  9-item Fear of Cancer Recurrence Inventory (FCRI-9, theoretical range: 0-36, where a higher score indicates a more pronounced fear of cancer recurrence). This scale is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.

SECONDARY OUTCOMES:
Health anxiety | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  14-item Health Anxiety Inventory (HAI-14, theoretical range: 0-42, where a higher score indicates more health anxiety). This scale is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Somatic symptom burden | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  Somatic Symptom Scale 8 (SSS-8, theoretical range: 0-32, where a higher score indicates a higher somatic symptom burden). Exploratory secondary analyses will be based on individual items, each scored 0-4. This scale is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Body image distress | Screening (within 6 months before treatment) to post-treatment assessment (immediately after treatment, completed within 90 days)
  Body Image Scale (BIS, theoretical range: 0-30, where a higher score indicates a higher level of body image distress)
Disability | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 90 days). Secondary analysis: from pre-treatment up to follow-up 12-months after treatment (completed within 90 days).
  12-item World Health Organization Disability Assessment Schedule 2.0 (WD2-12, theoretical range: 0-100, where a higher score indicates more disability). This scale is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Treatment credibility and patient expectancy of improvement | Week 2 of treatment
  Credibility/Expectancy scale (C/E scale, theoretical range: 0-50, where a higher score indicates higher credibility/expectancy)
Relationship with the therapist (therapeutic alliance) | Week 2 of treatment
  Working Alliance Inventory (WAI, theoretical range: 6-42, where a higher score indicates a stronger therapeutic alliance)
Patient satisfaction with treatment | Post-treatment assessment (immediately after treatment, completed within 90 days)
  8-item Client satisfaction questionnaire (CSQ-8, theoretical range: 8-32, where a higher score indicates higher satisfaction with treatment)
Adverse events | Post-treatment assessment (immediately after treatment, completed within 90 days)
  Brief questionnaire with three free-text items, each of which can be used to report an adverse event. For each adverse event, a rating is given of initial negative impact, and negative impact at post-treatment, on a scale from 0: "not at all", to 3: "very negatively". Reported primarily in terms of the number of participants reporting at least one adverse event.
Perceived negative effects of treatment | Post-treatment assessment (immediately after treatment, completed within 90 days)
  20-item Negative Effects Questionnaire (NEQ-20). This will be reported as the proportion of endorsed items in the following subdomains: increase in symptoms, perceived insufficient quality of treatment, dependency, stigma, and hopelessness.
Lifestyle behaviors | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 90 days).
  Lifestyle Behaviors Questionnaire (LBQ). The LBQ comprises 11 items that cover tobacco use, alcohol use, physical activity and diet. Dichotomous risky lifestyle behavior variables will be derived from the LBQ in terms of: "At least one unhealthy lifestyle behavior", "Daily smoking", "Binge drinking more than once a month OR more than 9/14 (w/m) glasses/week", "Insufficient physical activity, less than 150 minutes/week", and "Notably unhealthy dietary habits (diet index 0-4)". Risky lifestyle behavior will be defined as daily smoking, binge drinking of 4/5 (women/men) drinks at one occasion more than once a month and/or more than 9/14 (women/men) standard glasses of alcohol weekly, insufficient physical activity (<150 minutes/week) or significantly unhealthy diet habits (a score of 0-4 on a diet index in the questionnaire, ranging from 0-12).

OTHER OUTCOMES:
Process and target variables: Behavioral activation | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 90 days), and at follow-up 6 and 12 months after treatment (each completed within 90 days).
  3-item Behavioral Activation for Depression Scale - ACtivation subscale (BADS-AC-3, theoretical range: 0-18, where a higher score indicates a higher level of behavioral activation). This scale is also administered at screening (within 6 months before treatment), used to inform the eligibility assessment and to describe the sample.
Process and target variables: Symptom preoccupation | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 90 days), and at follow-up 6 and 12 months after treatment (each completed within 90 days).
  Symptom Preoccupation Scale (preliminary scale). A higher score indicates higher degree of preoccupation with symptoms. This is to be regarded as an an item pool, and the scale is is under development, which means that the total range cannot be preregistered.
Process and target variables: Physical activity | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 90 days), and at follow-up 6 and 12 months after treatment (each completed within 90 days).
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ, theoretical range 0-99, where a higher score indicates a higher level of physical activity). If necessary for statistical modeling, the GSLTPAQ will be dichotomized to indicate active (≥24) vs. insufficiently active (<24).
Process and target variables: Health-related self-efficacy | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 90 days), and at follow-up 6 and 12 months after treatment (each completed within 90 days).
  Based loosely on the Arthritis Self-efficacy Scale. Theoretical range of 0-60, where a higher score indicates a higher level of general health-related self-efficacy.
Basis for cost-effectiveness analysis: Utility (health-related quality of life) | Pre-treatment assessment (within 2 weeks before treatment), post-treatment assessment (immediately after treatment, completed within 90 days), 6 months after treatment (completed within 90 days), 12 months after treatment (completed within 90 days).
  EuroQol 5D (EQ-5D). Theoretical range: 0-1, i.e., scored as utility for the purpose of calculating quality-adjusted life years for health economic analysis. A higher utility score indicates a higher health-related quality of life.
Basis for cost-effectiveness analysis: Resource use (medical costs and productivity losses) | Pre-treatment assessment (within 2 weeks before treatment), post-treatment assessment (immediately after treatment, completed within 90 days), 6 months after treatment (completed within 90 days), 12 months after treatment (completed within 90 days).
  Trimbos Institute and Institute of Medical Technology Questionnaire for Costs Associated with Psychiatric Illness (TIC-P). This instrument is scored in terms of resource use for the purpose of calculating societal costs for health economic analysis.
Process and target variables: Health anxiety behaviors | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 90 days)
  Health Anxiety Behavior Inventory (HABI, scored as four subscales of "bodily preoccupation and checking", "information- and reassurance-seeking", "prevention and planning" and "overt avoidance"; each with a theoretical range of 0-9 where a higher score indicates a higher level of health anxiety behaviors within each respective subdomain)
Screening only: Alcohol use | Screening (within 6 months before treatment)
  Alcohol Use Disorders Identification Test (AUDIT, theoretical range: 0-40, where a higher score indicates more problematic alcohol use). This scale is administered to inform the eligibility assessment and describe the sample only.
Screening only: Substance use | Screening (within 6 months before treatment)
  Drug Use Disorders Identification Test (DUDIT, theoretical range: 0-44, where a higher score indicates more problematic substance use). This scale is administered to inform the eligibility assessment and describe the sample only.

CONTACTS AND LOCATIONS:
Overall Officials: Erland Axelsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this pilot study fall under Swedish and European Union data protection and privacy legislation and can therefore not be share in their entirety. Reasonable requests may be directed to the corresponding author, and will be considered on a case-by-case basis.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Original study protocol (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT06046586/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Amendments to the study protocol (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT06046586/SAP_001.pdf